CLINICAL TRIAL: NCT04582760
Title: Clinical Effect of Early Mobilization in Patients with Acute Respiratory Failure or Sepsis Requiring Mechanical Ventilation (Multicenter Randomized Controlled Trial by the Korean ICU Early Mobilization Network)
Brief Title: Early Mobilization in Ventilated SEpsis & Acute Respiratory Failure Study
Acronym: EVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Korea Health Industry Development Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019-11-143; HC19C0226 (Other: Korea Health Industry Development Institute)
Record Dates: First submitted 2020-07-22; First posted 2020-10-12 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Early Mobility; Critically Ill
Keywords: early mobility; Sepsis; Acute respiratory failure; Intensive care unit
MeSH Terms: conditions — Critical Illness; Sepsis | interventions — Early Ambulation; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- early mobilization Arm (Experimental): In addition to conventional bedside physical therapy, the mobilization program will be administered for 30 mins per session, two sessions per day, 7 days per week, until the patients are discharged from the ICU.
  Interventions: Other: early mobilization
- non-early mobilization Arm (No Intervention): Conventional bedside physical therapy will be administered for 30 mins per session, one session per day, 5 days per week (only on working days), until the patients are discharged from the ICU.

INTERVENTIONS:
Other: early mobilization — In patients who require mechanical ventilation for acute respiratory failure or sepsis (non-malignant tumor patients), early mobilization will be performed in addition to conventional bedside physical therapy, for 30 mins per session, two sessions per day, 7 days per week until the patients are discharged from the ICU.
  Other Names: physical therapy
  Arms: early mobilization Arm

SUMMARY:
Early mobilization in Ventilated sEpsis & acute Respiratory failure Study: EVER Study

DETAILED DESCRIPTION:
This is a multicenter, randomized, assessor-blinded study aiming to investigate the clinical effects of early mobilization in the ICU versus only conventional intensive care for improving physical function after ICU discharge, and after hospital discharge, in patients undergoing mechanical ventilation for acute respiratory failure or sepsis.

Recently, several studies on rehabilitation treatment for patients in intensive care have reported that rehabilitation treatment is safe for patients with ventilators, elderly patients, and patients receiving continuous renal replacement therapy (CRRT) or extracorporeal membrane oxygenation (ECMO). In the United States and Europe, evidence of the stability and clinical outcomes of physical and occupational rehabilitation in the ICU have already been established. In contrast, there is a lack of cost analysis and health and sociological grounds for intensive care rehabilitation in Korea. Therefore, there is an urgent need to evaluate the clinical effects of early rehabilitation, starting on the very first day in the ICU, in patients with acute respiratory failure and sepsis, requiring mechanical ventilation.

The clinical study plan of the current study is as follows. In ICU patients undergoing mechanical ventilation for acute respiratory failure or sepsis, the clinical effects of early mobilization on improving physical function will be assessed using FSS-ICU at discharge from the ICU and discharge from the hospital, and compared to those who did not receive early mobilization.

ELIGIBILITY:
Inclusion Criteria:You can participate in this clinical trial only if you meet all of the following criteria within 48 hours of ICU hospitalization.

* Those who voluntarily consent to participate in this clinical trial
* Those who are over the age of 18 years
* Patients who require mechanical ventilation for acute respiratory failure and sepsis (non-malignant tumor patients; excluding non-invasive mechanical ventilation and high-flow oxygen therapy)
* Patients with a Clinical Frailty Scale score of 1-4 points (physical condition prior to entering the ICU)
* Patients whose mechanical ventilation treatment is expected to last for more than 48 hours (evaluated at the time of study enrollment). However, if the patient has already begun mechanical ventilation treatment at another hospital, the time of airway intubation serves as the reference point. If it is difficult to confirm the exact time, the time of hospitalization is used as the reference point.

Exclusion Criteria:

* Patients with brain damage, psychiatric illness, or cognitive impairment making evaluation difficult
* Patients who are contraindicated for mobilization (active bleeding, deep vein thrombosis, increased brain pressure, open abdomen, iliac fracture, etc.
* Patients who do not meet the screening criteria for mobilization (however, if the ICU rehabilitation multidisciplinary team determines that mobilization can be started even if the patient does not meet the screening criteria below, the patient can be included in the study) A. Patients with a Richmond Agitation Sedation Scale (RASS) score less than -2 or greater than +2 B. Patients who have at least one of PEEP ≥ 10cmH2O, FiO2 ≥ 0.6, SpO2 < 90%, respiratory rate ≥ 35/min C. Patients who have at least one of systolic blood pressure <90 mmHg or> 200 mmHg, average arterial pressure> 110 mmHg or <65 mmHg, pulse rate> 130/min or <60/min or newly developed arrhythmia, or currently increasing the dose of inotropic agents.
* Patients who are pregnant
* Prisoners
* Patients with limitations in treatments (e.g., a declaration relating to life-sustaining treatment; or, if the patient is expected to die during hospitalization, if life-sustaining treatment is expected to be discontinued, or if the investigator expects a high probability of mortality (>50%))
* Patients who have already undergone mechanical ventilation treatment for more than 72 hours (if the patient is re-intubated within 36 hours after airway intubation, the treatment time is calculated as the continued mechanical ventilation time. If the total mechanical ventilation time is within 72 hours, the patient can be registered for the study)
* Patients who take neuromuscular blockers
* Patients whose physical function is impaired due to brain or spinal cord diseases
* Patients who weigh over 100kg
* Patients who maintain airway intubation and mechanical ventilation only to maintain airway hygiene
* Post-cardiac pulmonary resuscitation patients
* Those who are unsuitable for participation in the clinical trial due to other reasons including the results of clinical laboratory tests, according to the judgment of one of the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
FSS-ICU | Within 24 hours of ICU discharge
  Functional Status Score for the Intensive Care Unit Each task is evaluated using an eight-point ordinal scale ranging from 0 (unable to perform) to 7 (complete independence).The total score ranges from 0-35, with higher scores indicating better physical functioning.

SECONDARY OUTCOMES:
Length of ICU stay | Within 1 month of ICU discharge
  duration of hospitalization in ICU
Length of hospital stay | Wihin 1 month of hospital discharge
  duration of hospitalization
Mechanical ventilation treatment | Within 24 hours of ICU discharge
  Duration of mechanical ventilation treatment (28-day ventilator-free days)
Delirium-free duration | Within 24 hours of ICU discharge
  Delirium-free duration (28-day delirium-free days)
FSS-ICU | Wihin 24 hours of hospital discharge
  Functional Status Score for Intensive Care Unit(FSS-ICU)
MRC sum score | Wihin 24 hours of ICU discharge and hospital discharge
  Medical Research Council sum score (0-60;0-23,severe muscle weakness;24-35,moderate;36-47,mild)
Handgrip dynamometry | Wihin 24 hours of ICU discharge and hospital discharge
  Handgrip dynamometry
TUG | Wihin 24 hours of hospital discharge
  Timed Up and Go Test (TUG)
30s CSS | Wihin 24 hours of hospital discharge
  30s chair sit and stand (30s CSS)
CPAx-respiratory function | Wihin 24 hours of ICU discharge and hospital discharge
  The Chelsea Critical Care Physical Assessment Tool Respiratory function: Level 0-5 Level 0, complete ventilator dependence. Mandatory breaths only. May be fully sedated/paralised; Level 1, Ventilator dependence. Mandatory breaths with some spontaneous effort; Level 2, Spontaneously breathing with continuous invasive or non-invasive ventilatory support; Level 3, Spontaneouslu breathing with intermittent invasive or non-invasive ventilatory support or continuous high flow oxygen (>15L);Level 4, Receiving standard oxygen therapy (<15L);Level 5, Self-ventilating with no oxygen therapy
Health Care Costs | 1 year after discharged from the hospital
  Comparison of Health Care Costs
Use of Health Care Services | 1 year after discharged from the hospital
  Differences in the Use of Health Care Services
PICS surveys | 1 month, 3 months, 6 months, 12 months of hospital discharge
  Post Intensive Care Syndrome(PICS) surveys

CONTACTS AND LOCATIONS:
Overall Officials: GeeYoung Suh, MD PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: outcome instruments — https://www.improvelto.com/instruments/